CLINICAL TRIAL: NCT04545463
Title: Validation Study of the Effects of FIBRACEP Supplementation on the Lipid Profile
Brief Title: Hypocholesterolemic Effect of Fibracep
Acronym: FIBRACEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat de Lleida (Other)
Responsible Party: Principal Investigator, José Serrano, Principal Investigator, Universitat de Lleida
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CEIC-1534
Record Dates: First submitted 2020-09-02; First posted 2020-09-11 (Actual); Last update posted 2020-09-11 (Actual); Status verified 2020-09

CONDITIONS: Hypercholesterolemia
Keywords: Fiber; Cholesterol
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Insoluble Fibre (Active Comparator): Cookies with insoluble fibre (wheat bran)
  Interventions: Dietary Supplement: INSOLUBLE
- Soluble Fibre (Active Comparator): Cookies with soluble fibre (Psyllium plantago)
  Interventions: Dietary Supplement: SOLUBLE
- FIBRACEP (Experimental): Cookies with FIBRACEP
  Interventions: Dietary Supplement: FIBRACEP

INTERVENTIONS:
Dietary Supplement: FIBRACEP — A total intake of 7 g/day of FIBRACEP (provided in 6 cookies of 15 g/each) during two months
  Other Names: Onion fiber
  Arms: FIBRACEP
Dietary Supplement: INSOLUBLE — A total intake of 7 g/day of wheat bran (provided in 6 cookies of 15 g/each) during two months
  Other Names: Insoluble fibre from wheat bran
  Arms: Insoluble Fibre
Dietary Supplement: SOLUBLE — A total intake of 7 g/day of psyllium plantago (provided in 6 cookies of 15g/each) during two months
  Other Names: Soluble fibre from Psyllium plantago
  Arms: Soluble Fibre

SUMMARY:
FIBRACEP is an onion based fiber that has demonstrated in vitro and in animal models the capacity to increase HDL cholesterol levels as well to improve other lipid profile species. This intervention aims to demonstrate FIBRACEP's blood lipid profile improvement effect. For that purpose, hypercholesterolemic subjects will be recruited and given a daily dose of 7 g of FIBRACEP for two months. Changes in blood lipid profile will be the end-point of the study.

ELIGIBILITY:
Inclusion Criteria:

* Total cholesterol levels above 200 mg/dL, observed in at least 3 different days
* Body mass index between 25 and 35 (Overweight and obesity type 1 diagnosis)

Exclusion Criteria:

* Type 1 and Type 2 Diabetes
* Allergy to any compound described in FIBRACEP

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2016-05-01 (Actual); Study Completion 2016-05-01 (Actual)

PRIMARY OUTCOMES:
Blood HDL-cholesterol | 2 months
  Cholesterol content in HDL lipoproteins determined by nuclear magnetic resonance

SECONDARY OUTCOMES:
Blood lipid profile | 2 months
  Cholesterol content in LDL, VLDL (Very low-density lipoproteins) density and IDL lipoproteins determined by NMR
Blood lipoprotein number | 2 months
  Number of lipoproteins determined by nuclear magnetic resonance
Blood lipoprotein size | 2 months
  The average size of each lipoprotein specie (HDL, LDL, VLDL, IDL) determined by nuclear magnetic resonance

CONTACTS AND LOCATIONS:
Locations (1):
- José Serrano Casasola, Lleida, Spain

IPD SHARING:
Plan to Share IPD: Yes
By request to Principal Investigator
Supporting Information: Study Protocol, SAP, CSR
Time Frame: January 2021, for 2 years.
Access Criteria: By e-mail to Principal Investigator, who will decide to share the data if fulfill research purposes.